CLINICAL TRIAL: NCT05251467
Title: A Comprehensive Approach To Relief Of Digestive Symptoms In Cystic Fibrosis: CARDS-CF
Acronym: CARDS-CF
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); Royal Brompton & Harefield NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Sponsor
Other Study IDs: 21CS025
Record Dates: First submitted 2022-02-04; First posted 2022-02-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cystic Fibrosis; Digestive System Disease; Genetic Disease; Respiratory Tract Diseases; Lung Diseases; Pancreatic Disease
Keywords: Patient reported outcome measure (PROM); Gastrointestinal symptom burden; Symptom score; Gut; Abdomen
MeSH Terms: conditions — Cystic Fibrosis; Digestive System Diseases; Genetic Diseases, Inborn; Respiratory Tract Diseases; Lung Diseases; Pancreatic Diseases | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with CF age 12 years and over: Participants will be identified through one of the 6 participating UK CF centres as well as recruiting via social media. Participants outside the 6 listed CF centres as well as outside the UK are also eligible.
  Interventions: Other: Focus group; Other: Patient interview (n = approximately 10); Other: Questionnaire (n = 180); Device: Testing of the pilot PROM in a smartphone app (n = 150)

INTERVENTIONS:
Other: Focus group — Focus group to confirm PROM conceptual framework
Other: Patient interview (n = approximately 10) — Patient interviews to refine possible questions for the PROM
Other: Questionnaire (n = 180) — Online questionnaire to evaluate the proposed questions as part of PROM development in a larger population
Device: Testing of the pilot PROM in a smartphone app (n = 150) — Daily testing of the pilot PROM in a smartphone app for 2 weeks

SUMMARY:
Development of a new patient reported outcome measure (PROM) that will measure the daily burden of gastrointestinal symptoms over the previous 24 hour period for people with cystic fibrosis.

DETAILED DESCRIPTION:
Development of a Patient Reported Outcome Measure (PROM) in line with FDA guidance. The PROM is intended for daily use to measure the symptom burden of gastrointestinal symptoms for people with CF over the last 24 hours.

* Development of the initial conceptual framework underpinning the PROM and confirmed through a patient focus group.
* Primary item (question) generation for the PROM which will then be refined through a series of interviews with people with CF.
* Testing of the items through an online patient questionnaire for testing of frequency, burden and impact of the items.
* Piloting testing of the draft PROM daily for 2 weeks via smartphone app. The recall period of the PROM will be gastrointestinal symptom burden over the previous 24 hours.

Potential participant's will be identified through 6 UK CF care centres at Nottingham University Hospitals NHS Trust (paediatric and adult CF centres), Leeds Teaching Hospital NHS Trust, Manchester University NHS Foundation trust, Royal Brompton and Harefield NHS Foundation Trust and Kings College Hospital NHS Foundation Trust. In addition, recruitment for the survey and trialing the PROM on a smartphone app will also take place via social media and is therefore also open to people with CF from outside these CF centres.

ELIGIBILITY:
Inclusion Criteria:

* People with cystic fibrosis age 12 years and over
* Confirmed diagnosis of cystic fibrosis based on genotype or sweat chloride testing
* Capacity to consent, or to understand the requirements of the study where parental consent is required

Exclusion Criteria:

* < 12 years age
* Unable to give informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with cystic fibrosis age 12 years and over
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
To develop a new patient reported outcome measure (PROM) which will measure the daily gastrointestinal symptom burden for people with CF, with a recall period of 24 hours. | 2 years
  Development of a new PROM following FDA guidance which will measure the daily impact and burden of gastrointestinal symptoms for people with CF. The recall period will be the previous 24 hours. The name of the PROM will be decided as part of the development process. Question development will be iterative. Floor and ceiling effects for each of the questions will be assessed. The CFAbd score will be used to assess construct validity of the newly developed PROM. This will be completed alongside the PROM on days 1 and day 14.

SECONDARY OUTCOMES:
Measurement of adherence to daily data capture of the PROM through a smartphone app over a 2 week period | 2 years
  Adherence data - Percentage of completed PROM days over the 14 day period. Percentage of completed CFabd scores on days 1 and 14. This data will be collated through the research portal feedback facility in the app.
Attrition rate of participants | 2 years
  Attrition rate over the 2 weeks, define as people completing the app for two weeks (at least 10 out of 14 days) as a percentage of those initially who gave consent to take part and use the app.
Usability of the smartphone app | 2 years
  Usability of the app - participant feedback via the app on days 7 and 14 to include questions of ease of data entry on the app, whether they experience any technical issues with the app and whether questions are meaningful to participants. These questions will be developed as part of the PROM development process.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT05251467/Prot_SAP_002.pdf